CLINICAL TRIAL: NCT05253846
Title: Phase II Study of Short-course Radiotherapy Followed by Consolidation Chemotherapy With the Triplet FOLFOXIRI as Total Neoadjuvant Therapy for Locally Advanced Rectal Cancer: the ShorTrip Study
Brief Title: Short-course Radiotherapy Followed by Consolidation Chemotherapy. 2021-001206-29
Acronym: ShorTrip
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ShorTrip
Record Dates: First submitted 2022-01-17; First posted 2022-02-24 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Locally Advanced Rectal Cancer
Keywords: FOLFOXIRI; Locally advanced rectal cancer; Short-course radiotherapy; Total neoadjuvant strategy
MeSH Terms: interventions — Irinotecan; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SCRT--> FOLFOXIRI--> SURGERY (Experimental): SHORT-COURSE RT
  FOLFOXIRI
  * IRINOTECAN 165 mg/sqm iv over 60 minutes, day 1 followed by
  * OXALIPLATIN 85 mg/sqm iv over 2 hours, day 1 in two-way with
  * LEDERFOLIN 200 mg/sqm iv over 2 hours, day 1 followed by
  * 5-FLUOROURACIL 3200 mg/sqm 48 h-continuous infusion, starting on day 1. The chemotherapy treatment will be repeated every 2 weeks up to 8 cycles.
  Surgery with TME should be performed after 4 weeks after the last cycle of chemotherapy
  Interventions: Drug: Irinotecan; Drug: Oxaliplatin; Drug: Lederfolin; Drug: 5-Fluorouracil; Radiation: Short-course radiotherapy; Procedure: TME

INTERVENTIONS:
Drug: Irinotecan — chemotherapy treatment
Drug: Oxaliplatin — chemotherapy treatment
Drug: Lederfolin — treatment
Drug: 5-Fluorouracil — chemotherapy treatment
Radiation: Short-course radiotherapy — RT
Procedure: TME — surgery

SUMMARY:
The aim of the ShorTrip trail is to evaluate the activity and the safety of total neoadjuvant strategy with FOLFOXIRI as consolidation therapy preceded by short-course radiotherapy and followed by surgery in LARC patients.

DETAILED DESCRIPTION:
This is a prospective, open-label, multicentre, phase II single arm trial. Eligible patients with middle-high LARC will receive short-course radiotherapy followed by consolidation chemotherapy with FOLFOXIRI and surgery.

The primary objective of this trial is to evaluate the rate of complete pathologic response (pCR)

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to study procedures and to translational analyses;
* Age 18-70 years;
* Histologically proven diagnosis of rectal adenocarcinoma;
* Patients with locally advanced rectal cancer defined by the presence of at least one of the following features:

  * cN2 (defined as at least 4 positive lymphnodes at pelvic MRI)
  * cT4
  * tumor extending to within 1 mm of or beyond mesorectal fascia (i.e., circumferential radial margin threatened or involved)
  * cT3, N1
* Distal border of the tumour located between 5 and 12 cm from the anal verge (as measured by pelvic MRI);
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) ≤1;
* No evidence of metastatic disease by total body CT-scan;
* Available tumour samples at baseline (archival biopsy);
* Tumour amenable to curative resection (including pelvic exenteration);
* No history of invasive rectal malignancy, regardless of disease-free interval;
* No other rectal cancers (i.e., sarcoma, lymphoma, carcinoid, squamous cell carcinoma, or cloacogenic carcinoma) or synchronous colon cancer;
* No clear involvement of the pelvic side walls by imaging;
* Life expectancy of at least 5 years (excluding diagnosis of cancer);
* Hematopoietic function: absolute neutrophil count ≥ 1,500/mm3; platelet count

  ≥100,000/mm3; haemoglobin level ≥ 9 g/dL;
* Liver function: total bilirubin ≤ 1.5 times upper limit of normal (ULN); alkaline phosphatase ≤ 2 times ULN; AST ≤ 2 times ULN;
* Renal function: creatinine clearance > 50 mL/min or serum creatinine 1.5 x UNL; no renal disease that would preclude study treatment or follow-up;
* Women of childbearing potential must have a negative blood pregnancy test at the screening visit. For this trial, women of childbearing potential are defined as all women after puberty, unless they are postmenopausal for at least 12 months, are surgically sterile, or are sexually inactive. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy.

However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient; - Subjects and their partners must be willing to avoid pregnancy during the trial. Male subjects with female partners of childbearing potential and female subjects of childbearing potential must, therefore, be willing to use adequate contraception.

Contraception, starting during study screening visit throughout the study period up to 180 days after the last dose of chemotherapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject;

- Will and ability to comply with the protocol.

Exclusion Criteria:

* Previous history of malignancy within the last 5 years will be excluded with the exception of localized basal and squamous cell carcinoma or cervical cancer in situ;
* Patients with radiological evidence of distant metastases;
* Previous pelvic radiation therapy;
* Symptomatic peripheral neuropathy > 2 grade NCIC-CTG criteria;
* Previous treatment with fluoropyrimidine and/or oxaliplatin and/or irinotecan;
* Patient with complete dihydropyrimidine dehydrogenase (DPYD) deficiency (homozygous of the following DPYD polymorphisms: c1679GG, c1905+1AA, c2846TT);
* Treatment with any investigational drug within 30 days prior to enrolment or 2 investigational agent half-lives (whichever is longer);
* Active uncontrolled infections or other clinically relevant concomitant illness contraindicating chemotherapy administration;
* Clinically significant (e.g. active) cardiovascular disease for example cerebrovascular accidents (≤6 months), myocardial infarction (≤6 months), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure (CHF), serious cardiac arrhythmia requiring medication;
* Active inflammatory bowel disease (i.e., patients requiring current medical interventions or who are symptomatic);
* Partial or total colectomy;
* Pregnant or lactating women. Women of childbearing potential with either a positive or no pregnancy test at baseline. Sexually active males and females (of childbearing potential) unwilling to practice contraception during the study and until 180 days after the last trial treatment;
* Known hypersensitivity to fluorouracil, oxaliplatin or irinotecan;
* Psychiatric or addictive disorders, or other conditions that, in the opinion of the investigator, would preclude study participation;
* Active uncontrolled infections or other clinically relevant concomitant illness contraindicating chemotherapy administration;
* Withdrawal of the consent to take part to the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2025-01-05 (Actual); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
complete pathologic response (pCR) | 30 months
  Pathological complete response rate, defined as the percentage of patients, relative to the total of enrolled subjects, with the absence of residual tumour cells in the resected specimens. pCR will be assessed by tumour regression grade according to Dworak et al, at the histopathological exam

SECONDARY OUTCOMES:
Overall toxicity rate | 30 months
  Overall toxicity rate, defined as the percentage of patients, relative to the total of enrolled subjects, who receive radiotherapy and at least one cycle of chemotherapy, experiencing any adverse event, according the RTOGTC during SCRT, and according to National Cancer Institute Common Toxicity Criteria (version 5.0), during the consolidation chemotherapy
G3/4 toxicity rate | 30 months
  G3/4 toxicity rate, is defined as the percentage of patients, relative to the total of enrolled subjects, who receive radiotherapy and at least one cycle of chemotherapy, experiencing a specific adverse event of grade 3/4, according the RTOGTC during SCRT, and according to National Cancer Institute Common Toxicity Criteria (version 5.0), during the consolidation chemotherapy.
R0 Resection Rate | 30 months
  R0 Resection Rate is defined as the percentage of patients, relative to the total of enrolled subjects, undergoing R0 resection of primary tumour. R0 surgery is defined as microscopically margin-negative resection at the histopatological exam
Failure-free survival (FFS) | 7 years
  Failure-free survival (FFS) is defined as the time from enrollment to one of the following events: non-radical surgery (non R0/R1) of the primary tumour, intrapelvic recurrence after R0/1 resection of the primary tumour, distant relapse, second primary tumour or death from any cause, whichever occurred first. The determination of disease progression will be based on investigator-reported measurements. Patients who are alive without having one of the above events at the end of the study will be censored at their last radiological assessment
Overall Survival (OS) | 7 years
  Overall Survival (OS) is defined as the time from enrolment to death from any cause. For patients still alive at the time of analysis, the OS time will be censored on the last date the patients were known to be alive
Time to distant metastases | 7 years
  Time to distant metastases, is defined as the time from enrolment to the radiological evidence of distant metastases. The determination of the evidence of distant metastases will be based on investigator-reported measurements. Patients who are died or alive without having distant metastases at the end of the study will be censored at the date of death or their last radiological assessment, respectively
Time to locoregional failure | 7 years
  Time to locoregional failure is defined as the time from the enrolment to non-radical surgery of the primary tumour (non R0/R1 resection) or intrapelvic recurrence after R0/1 resection of the primary tumour. The determination of the intrapelvic recurrence will be based on investigator-reported assessment. Patients who are died or alive without having non-radical surgery or intrapelvic recurrence at the end of the study will be censored at the date of death or at their last radiological assessment
Clinical complete response (cCR) rate | 30 months
  Clinical complete response (cCR) rate, defined as the percentage of patients, relative to the total of enrolled subjects, with the absence of residual tumour (cT0cN0) at the radiological and endoscopic staging after neoadjuvant treatment.
Major pathological response (MPR) rate | 30 months
  Major pathological response (MPR) rate, defined as the percentage of patients, relative to the total enrolled subjects, achieving TRG1-2 sec Mandard or TRG3-4 sec Dworak at the histopathological exam
Surgical mortality | 30 months
  Surgical mortality, defined as the percentage of patients, relative to the total of enrolled subjects, experiencing death within 30 days after the surgery
Surgical morbidities | 30 months
  Surgical morbidities, defined as the percentage of patients, relative to the total of enrolled subjects, experiencing any post-operative complications within 30 days after the surgery
Quality of Life (QoL) | until 1 year after surgery
  Quality of Life, (QoL) assessed using the EORTC QLQ-C30, will be evaluate at specific time-points (baseline, after radiotherapy, and chemotherapy, after surgery and during follow-up) and will be assessed through descriptive summary statistics
Quality of Life (QoL) | until 1 year after surgery
  Quality of Life, (QoL) assessed using the EORTC QLQ-CR29, will be evaluate at specific time-points (baseline, after radiotherapy, and chemotherapy, after surgery and during follow-up) and will be assessed through descriptive summary statistics
Quality of Life (QoL) | until 1 year after surgery
  Quality of Life, (QoL) assessed using the EuroQol EQ-5D questionnaires, will be evaluate at specific time-points (baseline, after radiotherapy, and chemotherapy, after surgery and during follow-up) and will be assessed through descriptive summary statistics
Rectal Continence | until 180 days after the ileostomy closure surgery
  Rectal Continence, assessed using LARS scores, will be evaluate at specific time-points (baseline, after radiotherapy, and chemotherapy, after surgery and during follow-up) and will be assessed through descriptive summary statistics
Rectal Continence | until 180 days after the ileostomy closure surgery
  Rectal Continence, assessed using St. Mark Continence scores, will be evaluate at specific time-points (baseline, after radiotherapy, and chemotherapy, after surgery and during follow-up) and will be assessed through descriptive summary statistics

OTHER OUTCOMES:
Correlation of FFS and pCR with ctDNA status | 7 years
  Correlation of FFS and pCR with ctDNA status, assessed at prespecified timepoints during the study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Moretto, MD, Principal Investigator — Azienda Ospedaliero, Universitaria Pisana
Locations (1):
- U.O. Oncologia Medica 2 Universitaria - Azienda Ospedaliero-Universitaria Pisana Dipartimento di Ricerca Traslazionale e Nuove Tecnologie - University of Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No